CLINICAL TRIAL: NCT04492202
Title: Comparison of the Knowledge, Attitudes, and Practices Towards COVID-19 Between Different Healthcare Professionals
Brief Title: Knowledge, Attitudes, and Practices Towards COVID-19 Among Health Care Professionals Among Healthcare Professionals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Other Study IDs: 00010
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: COVID; Knowledge, Attitudes, Practice
Keywords: Health Care Professionals
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- First group: Physiotherapists will be included in this group.
  Interventions: Other: Survey
- Second group: Doctors will be included in this group.
  Interventions: Other: Survey
- Third group: Nurses will be included in this group.
  Interventions: Other: Survey
- Fourth group: Other health professionals will be included in this group.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The survey will be sent to health professionals via online link.

SUMMARY:
The aim of this study is to evaluate the knowledge level of healthcare professionals such as physicians, nurses, physiotherapists and nutritionist about published COVID-19 guidelines.

The listed healthcare workers are take part in the primary treatment of the Corona virus infected patients in hospitals. Therefore the knowledge of the world wide spreading Corona Virus and its effects for the human being is should be known for the effective treatment and for raising public awareness.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, nurses, physiotherapists and other healthcare professionals with clinical practical experience
* Actively working in the hospitals and in any health institution

Exclusion Criteria:

* Employees outside the health area
* Health professionals who do not work in any health institution
* Employees who do not have a bachelor's degree

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our planned study is physician, nurse, physiotherapist, etc. It is designed to measure the knowledge, attitudes and practices of all professionals working in the field of health.
  The study designed to measure the knowledge, attitudes and practices of all professionals such as physician, nurse, physiotherapist and nutritionist working in the field of medical and health sciences.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Questionnaire for the Evaluation of Knowledge, Attitude and Practise Levels of Healthcare Professionals for COVID-19 | 4 weeks
  The purpose of the knowledge, attitude and practise questionnaire; to measure the knowledge, attitude and skill levels of healthcare professionals against the COVID-19 virus. In addition, this study will demonstrate the change in the knowledge, attitudes and practise of different healthcare professionals regarding COVID-19. This questionnaire was developed by Istinye University Faculty of Health Science, Physiotherapy and Rehabilitation Department.

SECONDARY OUTCOMES:
Support Approach Survey for Patients in Recovery Stage after COVID-19 Diagnosis | 4 weeks
  This questionnaire has been used to evaluate the knowledge and guidance of healthcare professionals about which best approaches can be used to support patients who have had COVID-19 diagnosis and recovered. This questionnaire was developed by Istinye University Faculty of Health Science, Physiotherapy and Rehabilitation Department.

OTHER OUTCOMES:
Fear of COVID-19 Scale | 4 weeks
  The emergence of the COVID-19 and its consequences has led to fears, worries, and anxiety among individuals and health professionals worldwide. The Fear of COVID-19 Scale (FCV-19S) was developed to complement the clinical efforts in preventing the spread and treating of COVID-19 cases. We are going to evaluate the fear of COVID-19 in health professionals.